CLINICAL TRIAL: NCT06566742
Title: A Phase 2 Study Evaluating Olutasidenib in Patients With IDH1-mutated Clonal Cytopenia of Undetermined Significance and Lower-risk Myelodysplastic/Syndromes/Chronic Myelomonocytic Leukemia.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0509; NCI-2024-07045 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Clonal Cytopenia of Undetermined Significance
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — olutasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olutasidenib (Experimental): Participants will take capsules of olutasidenib 2 times each day while you are on study. Each dose should be taken about 12 hours apart at least 1 hour before or 2 hours after a meal.
  Interventions: Drug: Olutasidenib

INTERVENTIONS:
Drug: Olutasidenib — Given by PO

SUMMARY:
To learn if olutasidenib can help to control CCUS, MDS, and/or CMML. The safety of the drug will also be studied.

DETAILED DESCRIPTION:
Primary Objectives - To determine the response rate of olutasidenib monotherapy in patients with IDH1-mutated CCUS or lower-risk MDS/CMML

Secondary Objectives

* To evaluate the rates of transfusion independence, defined as the absence of transfusions over a period of at least 8 weeks
* To ascertain the safety and tolerability of olutasidenib monotherapy in these participants populations
* To determine survival and rates of leukemia transformation
* To analyze reduction in IDH1 clone size

Exploratory Objectives

- To investigate global gene expression profiles, DNA methylation profiles, and other potential prognostic markers to explore predictors of antitumor activity and/or resistance to treatment.

OUTLINE:

Patients receive olutasidenib orally (PO) twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with CCUS receive up to 18 months of olutasidenib. Patients with lower-risk MDS/CMML can receive olutasidenib until disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and bone marrow aspiration and biopsy on study.

After completion of study treatment, patients are followed up every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven CCUS or lower-risk MDS/CMML.

   1. CCUS is defined as the presence of cytopenia (absolute neutrophil count < 1.8 x 10^9/L, hemoglobin < 13 g/dL in males or < 12 g/dL in females, and/or platelets < 150 x 10^9/L) for at least 30 days that are otherwise unexplained and with no diagnostic hematopathologic features of myeloid neoplasms. Patients with known Duffy-null phenotype must have absolute neutrophil counts less than their lower limit of normal.
   2. Lower-risk MDS/CMML includes patients with International Prognostic Scoring System (IPSS) low- or intermediate-1-risk disease and Revised IPSS (IPSS-R) score ≤ 3.5 and Molecular IPSS (IPSS-M) very low-, low-, or moderate low-risk categories.
2. Patients must have a documented IDH1 mutation with variant allele frequency (VAF) ≥ 0.02.
3. Patients ≥ 18 years old.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
5. Bilirubin ≤ 2 times upper limit of normal (ULN) or ≤ 3 times ULN in patients with Gilbert Syndrome.
6. Aspartate transaminase (AST), alanine transaminase (ALT), and alkaline phosphatase ≤ 3 times ULN.
7. Acceptable renal function with serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance ≥ 50 mL/min (as assessed by Cockcroft-Gault, Modification of Diet in Renal Disease Formula [MDRD], or Chronic Kidney Disease Epidemiology [CKD-Epi] validated measures).
8. Negative serum or urine pregnancy test if female of childbearing potential.
9. For fertile men and women, agreement to use highly effective contraceptive methods for the duration of study participation and 90 days after the last dose of study medication. Appropriate highly effective method(s) of contraception include oral or injectable hormonal birth control, intrauterine device (IUD), and double barrier methods (for example a condom in combination with a spermicide).
10. Agreement for male patients not to donate sperm and for female patients of childbearing potential not to donate ova during the study and for 90 days after the final dose of study drug.
11. Ability and willingness to signed informed consent prior to beginning study and undergoing procedures.

Exclusion Criteria:

1. Patients unable to swallow oral medications, or patients with gastrointestinal conditions (e.g., malabsorption, resection, etc.) deemed by the Investigator to jeopardize intestinal absorption.
2. Patients with any concurrent uncontrolled clinically significant medical condition, including life-threatening severe infection or psychiatric illness, which could place the patient at unacceptable risk of study treatment.
3. Known active hepatitis B (hepatitis B virus [HBV]) or hepatitis C (hepatitis C virus [HCV]) or HIV infection.
4. Pregnant or nursing women or women of childbearing potential not using highly effective contraception; male patients not using highly effective contraception as defined in the inclusion criteria.
5. Subject with white blood cell count > 25 x10^9/L.

   * Note: hydroxyurea use is permitted to meet this criterion with no washout required.
6. Unwillingness or inability to comply with procedures either required in this protocol or considered standard of care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Chien, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org